CLINICAL TRIAL: NCT02181257
Title: Extracorporeal Photopheresis for the Management of Progressive Bronchiolitis Obliterans Syndrome in Medicare-Eligible Recipients of Lung Allografts
Brief Title: Extracorporeal Photopheresis for Medicare Recipients of Lung Allografts
Acronym: ECP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Centers for Medicare and Medicaid Services/ Coverage and Analysis Group (U.S. Federal Agency); Therakos, Inc (Unknown); The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201402035
Record Dates: First submitted 2014-07-01; First posted 2014-07-03 (Estimated); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Bronchiolitis Obliterans Syndrome (BOS)
Keywords: Bronchiolitis Obliterans Syndrome; Lung Transplantation; Extracorporeal Photopheresis; Methoxsalen; Chronic lung allograft dysfunction (CLAD)
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Photopheresis

STUDY DESIGN:
Intervention Model Description: REFRACTORY BOS - Participants are electronically assigned to either ECP Treatment or Observation (Standard Immunosuppression Therapy)
  NEW BOS Participants are randomized to ECP Treatment or Control (Standard Immunosuppression Therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Newly Diagnosed Bronchiolitis Obliterans (NEW BOS) (Other): Participants with NEW BOS will be randomized to Early Photopheresis Intervention (EPI) or Control (Standard of Care). EPI patients will receive 24 treatments in a 6-month period and may continue maintenance treatments. Twenty-two (22) NEW BOS participants were enrolled nationwide.
  The Control group will receive local Standard of Care for the management of BOS. Therapy will involve changes in immunosuppressive agents.
  Interventions: Combination Product: Extracorporeal Photopheresis (ECP)
- Refractory Bronchiolitis Obliterans Syndrome (REFRACTORY BOS) (Other): Participants with REFRACTORY BOS will be electronically assigned to either ECP treatment or Observation based on the participant's pre-enrollment Forced Expiratory Volume in 1 second (FEV1). Values from pulmonary function tests from the preceding 12 months will be entered into a web-based treatment allocation which will perform an automated calculation. Patients who have a statistically significant rate of decline within the preceding 6 months, and a derived protocol defined slope, will be assigned to the ECP Treatment arm. If a patient does not meet these criteria, the participant will be assigned to the Observation arm.
  Two hundred and fifty-eight (258) participants were enrolled with Refractory BOS nationwide.
  Interventions: Combination Product: Extracorporeal Photopheresis (ECP)
- Standard of Care Comparator Retrospective Chart review (Other): Data for the SOC comparator will be obtained via a retrospective data capture mechanism either medical chart review or electronic medical record query that meet all of the inclusion criteria and through an IRB approved waiver of consent. The SOC comparator data will be identical to the data collected for the Refractory BOS patients with the exception of inclusion of all spirometry values after transplant.
  Interventions: Other: No intervention in the SOC / Retrospective Chart review.

INTERVENTIONS:
Combination Product: Extracorporeal Photopheresis (ECP) — Procedure:
  ECP treatments will be performed using one of two Therakos systems. Both systems use the drug Methoxsalen
  Arms: Newly Diagnosed Bronchiolitis Obliterans (NEW BOS); Refractory Bronchiolitis Obliterans Syndrome (REFRACTORY BOS)
Other: No intervention in the SOC / Retrospective Chart review. — SOC Retrospective chart review similar to a control group
  Arms: Standard of Care Comparator Retrospective Chart review

SUMMARY:
The primary aims of this study is to determine the efficacy and tolerability of Extracorporeal Photopheresis (ECP) for the treatment of either Refractory Bronchiolitis Obliterans Syndrome (BOS) patients (258 at cessation of enrollment April 7, 2022) or Newly Diagnosed (22 as of enrollment Hold February 2022) Bronchiolitis Obliterans Syndrome patients after lung transplantation. In compliance with the Centers for Medicare and Medicaid Services' (CMS) Coverage with Evidence Development (CED) decision, the study will collect specified demographic, comorbidity, treatment, and outcome data exclusively for Medicare beneficiaries who are treated with ECP for either refractory or New BOS.

DETAILED DESCRIPTION:
Lung transplantation has become the treatment of choice for selected patients with end-stage lung disease. Long-term survival after transplantation remains disappointing. Chronic rejection in the form of bronchiolitis obliterans syndrome (BOS) has emerged as the leading obstacle to better long-term outcomes, and is the leading cause of death beyond the first year after transplantation. This disorder is a fibroproliferative scarring process that involves the narrowing of the airway lumen and ultimately complete luminal obliteration. Physiologically and clinically, this luminal narrowing results in airflow limitation and breathlessness. Histologic confirmation of BOS is difficult with bronchoscopy obtained lung biopsies because of the patchy distribution of the disorder and inadequate sampling of small airways with transbronchial lung biopsies. As a result, BOS is diagnosed and staged by the decline in Forced Expiratory Volume in 1 Second (FEV1) measurement from a pulmonary function test.

In general, BOS is treated by intensifying the immunosuppressive regimen. The specific approach is variable from center to center, but typically includes optimizing the maintenance immunosuppressive regimen to include tacrolimus and mycophenolate mofetil, high-dose steroids, and a course of anti-thymocyte globulin. Despite treatment, most patients continue to show progressive decline in lung function resulting in worsening functional status, quality of life, and ultimately graft failure and death.

Extracorporeal photopheresis (ECP) has been used at some centers as a salvage treatment for progressive BOS. ECP involves separating the patient's blood into a leukocyte-enriched component (buffy coat) and a leukocyte-depleted component. The buffy coat is then photosensitized with 8-methoxypsoralen and treated with ultraviolet light within a photosensitization chamber, resulting in leukocyte apoptosis. Although the exact mechanism of action of ECP is unclear, re-infusion of this apoptotic leukocyte population into the patient's circulation is thought to result in alterations in antigen presenting cells, cytokine profiles, and the expansion of regulatory T cells.

On May 2, 2012, the Centers for Medicare & Medicaid Services issued a Decision Memo stating that ECP is covered for Medicare beneficiaries for the treatment of BOS following lung allograft transplantation only when the procedure is provided under a clinical research study.

This study looks at (1) Early detection of refractory BOS using a standardized, more frequent spirometry monitoring approach (i.e., defined as using frequent laboratory based spirometry every 4-8 weeks) and (2) Early implementation of ECP in both participants with early stage refractory BOS and also as first line therapy in a subset of participants at the initial diagnosis of BOS, in the context of a new randomized controlled trial.

The study will look at whether certain coexisting disease states or patient-related demographic, functional, treatment-related or diagnostic variables (e.g. extent or statistical significance of the rate of pre-ECP FEV1 decline) might prove to have predictive value in identifying subsets of BOS patients that are likely, or unlikely, to experience reduced rate of decline or stabilization in FEV1 following ECP treatment. Therefore this study will look to enroll a large series of patients from multiple U.S. centers to confirm that ECP significantly reduces the rate of FEV1 decline in BOS patients refractory to standard immunosuppressive drug therapy, and to capture and assess specified patient demographic, treatment-related, diagnostic, functional and co-morbidity-related variables that may predict outcomes after ECP therapy. Enrollment is now complete and ended April 6, 2002. Patients are now in follow-up and will be followed no later than the end of the study December 2028.

This study includes a randomized controlled trial that will compare outcomes in patients with newly diagnosed BOS who receive either conventional (i.e., that involves the standard of care at the respective enrolling center) or ECP for first line management of New BOS. The randomized controlled trial component of the study will enable evaluation of potential survival and quality of life benefits of early treatment of BOS with first-line ECP. The randomized control trial was placed on hold in February of 2022. Twenty-two patients were enrolled study wide. Patients are now in follow-up and will be followed no later than the end of the study December 2028.

Subjects with Refractory BOS who agreed to participate in the study were informed of the following: to limit the use (and attendant risks) of ECP therapy to those patients who are most likely to benefit, their eligibility to receive ECP within the study will be determined by the study team's analysis of their pre-enrollment pulmonary function testing along with input from their physician.

Subjects with Newly-Diagnosed BOS who agreed to participate in the study were informed that they will be randomly assigned to either a control group (Control) who will receive the local Standard of Care for management of their BOS or to an Early Photopheresis Intervention (EPI) group who will receive ECP as first line management of BOS.

The protocol states specific inclusion and exclusion criteria for both the Refractory BOS participant and the newly diagnosed BOS participant. Once eligibility is confirmed and the patient has provided informed consent, all FEV1 measurements captured within the 12 months prior to enrollment will be entered in the electronic database. Based on the slope of the FEV1 decline over time and achievement of a statistically significant rate of decline in lung function in the FEV1 the Refractory BOS participant will be electronically assigned to either ECP treatment or Observation. The newly diagnosed BOS participant will be randomized to either ECP treatment and standard immunosuppression therapy or Control treatment which is Standard immunosuppression Therapy alone.

The participant will be assigned a unique identification number created from the electronic data base. The patient demographics, co-morbidities, medical history including date of lung transplantation, underlying disease necessitating lung transplantation, vital signs, height, weight, and current immunosuppression regimen will be entered at baseline. A Quality of Life Questionnaire will be asked at baseline and every 3 months the first year and then annually. A pulmonary function test will be captured every 30 days for the first year on all patients except the Refractory BOS participant assigned to Observation. Pulmonary function tests will be captured every 30 days for the first six months for the Observation patient. Following the first six months, the timing of pulmonary function testing must be every 3 months at the very least to maintain eligibility for ECP Treatment. Certain de-identified source documents will be required and verified on all forms electronically submitted. Data points will be verified against de-identified source by the Data Coordinating Center. The online data entry portal and study database will contain a mechanism to a) clearly denote the status of each submitted Case Report Form, including whether the case report form is complete; b) list the source documentation needed c) indicate if the site staff member and investigator have attested to the validity of the data on the Case Report Form; and d) indicate if the Data Coordinating Center has verified the accuracy of key elements of the study data and what data queries remain. This centralized monitoring will complement our remote monitoring visits during COVID. For most sites an initial remote site monitoring visit will occur after the first three patients are enrolled to ensure that the site personnel understand study processes and expectations, and to permit early completion of additional training to address any deficiencies. Should remote or on-site monitoring reveal areas of particular deficiency or concern, the monitoring plan will be adjusted to focus on those particular areas for the site. In general, sites and patients affiliated with a major violation will be monitored with greater completeness. Sites deemed to be largely compliant with the protocol and regulatory requirements based upon the initial monitoring visit are expected to have subsequent visits performed at a reduced level of frequency. Overall, the study team will seek to optimize resource use by focusing on the most critical data elements that may impact subject safety and/or data quality and integrity.

Participants who receive ECP treatment will receive 24 treatments over the 6-month period following enrollment.

Allowed Treatment for Refractory BOS patients in the Observation will be ordered at the physicians discretion.

Treatment for the Newly Diagnosed BOS patients in the Control Arm of the randomized control trial will be dictated by the standard of care within each enrolling institution and will involve changes in immunosuppressive agents. These patients will not be eligible to receive ECP treatment.

Other than ECP, no other interventions for BOS will be used except for Azithromycin for patients in the randomized Early Photopheresis Intervention arm.

An improvement in the FEV1 measurement taken from the pulmonary function test will be used to assess the success or the benefit of the ECP treatment. Patients will have spirometry the first week of therapy, which is repeated every 30 days for the first year, and then annually in the Refractory BOS cohort assigned to ECP treatment. Patient's will have spirometry the first week of therapy, and repeated every 30 days for the first year, and then every 2 months in the NEW BOS cohort. All patients will be followed no later than December 2028. There were considerations for crossover built into the early versions of the protocol.

Statistical Methods. The primary outcome in the RCT or New BOS will look at cumulative all cause mortality and the rate of decline of lung function: A 25% or greater difference in the percentage of patients within each of the two arms (Control vs Early photopheresis Intervention(EPI) who achieve a clinical response as defined as 50% or greater reduction in the rate of FEV1 decline as assessed by comparing the average rate of FEV1 decline over the 6 months prior to ECP against the average rate of FEV1 decline over the 12 months following randomization.

The primary endpoint in the Refractory BOS registry involves a change in the rate of FEV1 decline assessed by comparing the average rate of FEV1 decline over the 6 months prior to ECP against the average rate of FEV1 decline over the 12 months following initiation of ECP. A clinical response will be determined using FEV1 as the primary endpoint and will be defined as a 50% or greater reduction in the rate of decline of FEV1 assessed by comparing the average rate of FEV1 decline over the 6 months prior to ECP against the average rate of FEV1 decline over the 12 months following initiation of ECP. A clinical response will be defined as a 50% or greater reduction in the rate of decline of FEV1 before and after the ECP. The second primary endpoint will include all cause and CLAD related mortality.

The participants will be followed until their death but no later than December 2028 and the following data will be collected annually after the first year: Spirometry results, the number of maintenance Extracorporeal Photopheresis treatments performed and Quality Of Life surveys will be tabulated.

In parallel, data will be collected retrospectively from up to 250 lung transplant recipients (through an IRB approved waiver of consent) who developed NEW BOS and were treated with standard of care (SOC) therapy and did not receive ECP treatment. The addition of a propensity matched standard of care BOS Cohort may promote a more robust assessment of the potential clinical impact of ECP.

ELIGIBILITY:
INCLUSION Criteria for REFRACTORY BOS

1. Age (18 years old or older).
2. Medicare-eligible status
3. Lung transplant recipient (combined organ transplant recipients, e.g. heart-lung or liver-lung or lung re- transplantation recipients are eligible).
4. Patients with a diagnosis of BOS using at least two laboratory based FEV1 values obtained at least three weeks apart that are both at least 20% lower than baseline FEV1 using the International Society for Heart and Lung Transplantation (ISHLT) definition (The average of the two highest FEV1 measurements obtained at least 3 weeks apart after transplantation). The date of Diagnosis of New BOS is the first date of the two FEV1s that were used for the BOS diagnosis.
5. Refractory BOS defined as ongoing decline in FEV1 despite at least one of the following treatments:

   azithromycin, high-dose steroid, anti-thymocyte globulin, total lymphoid irradiation, sirolimus, or everolimus.
6. At minimum five recorded FEV1 measurements obtained at intervals of at least two weeks apart, over the 9 months preceding study enrollment, of which one FEV1 must be within two weeks prior to enrollment.
7. History of frequent spirometry monitoring defined as having had regular FEV1 measurements within the context of either of the following two options: (1) During the preceding four months prior to enrollment with no time interval between FEV1 measurements that exceeds 8 weeks. (2) During the preceding six months prior to enrollment with no time interval between FEV1 measurements that exceeds 12 weeks.
8. A documented clinical assessment including a physical assessment and Complete Blood Count (CBC) with White Blood Cell Count (WBC) within two weeks prior to enrollment.

INCLUSION criteria for NEWLY Diagnosed BOS

1. Age (18 years old or older)
2. Medicare-eligible status.
3. Lung transplant recipient (combined organ transplant recipients, e.g. heart-lung or liver-lung, lung re-transplantation recipients, are eligible).
4. History of close FEV1 monitoring prior to diagnosis of new BOS defined as having had either of the two monitoring approaches:

<!-- -->

1. Frequent laboratory based spirometry defined as having had regular FEV1 measurements within the context of either of the following two options: A. During the preceding six months prior to diagnosis of new BOS with no time interval between FEV1 measurements that exceeds 8 weeks. (Participants must be at least 6 months post transplant) B. During the preceding nine months prior to diagnosis of new BOS with no time interval between FEV1 measurements that exceeds 12 weeks (Participants must be at least 9 months post- transplant)
2. Frequent Home Spirometry through the separate IRB approved Standardized Home Spirometry Method sub-protocol. 5.Diagnosis of new BOS (i.e., "new BOS" is defined as within nine weeks of enrollment) based on laboratory-based spirometric FEV1 measurements obtained on at least two separate occasions (i.e., at least 3 weeks apart) that have declined by more than 20% from post-transplant baseline values (i.e., using ISHLT definition). The date of Diagnosis of New BOS is the first date of the two FEV1s that were used for the BOS diagnosis. Inherent to the diagnosis of new BOS is the exclusion of other potential causes of allograft dysfunction such as acute rejection, respiratory tract infection, and airway anastomotic complications. Thus, sites are encouraged to conduct appropriate evaluation for declining allograft function including bronchoscopy with bronchoalveolar lavage (BAL) and lung biopsies if clinically appropriate to exclude other potential causes of allograft dysfunction. 6. Achievement of a statistically significant rate of decline in lung function (FEV1) at the diagnosis of new BOS per the criteria in

Section 3.6 as assessed by the following criteria:

1. For patients who are monitored with laboratory based spirometry, at least five recorded FEV1 measurements obtained at intervals of at least two weeks apart, over either the 6 or 9 (i.e., depending on the frequency of spirometry testing) months preceding study enrollment accompanied by a statistically significant (p<0.05) rate of decline of FEV1 that exceeds 30 mL/month; or
2. For patients who are monitored with home Spirometry, 4-6 recorded home spirometry FEV1 measurements obtained one week apart, over the 4-6 weeks prior to a confirmed FEV1 variance (i.e., the date of the second of two consecutive FEV1 values below the patient's normal range) along with 4-6 recorded weekly FEV1 measurements obtained after a confirmed variance accompanied by a statistically significant (p<0.05) rate of de-cline of FEV1 that exceeds 30 mL/month 7. Documented clinical assessment including a physical assessment and a CBC with WBC within two weeks prior to enrollment.

EXCLUSION Criteria (Subjects meeting any one of these criteria will be excluded)

1. Current participation in another clinical treatment trial with an investigational agent used to manage BOS before or after enrollment.
2. Any condition that may interfere with the subject's ability to perform pulmonary function testing.
3. Known allergy or hypersensitivity to pharmacologic agents used during ECP
4. Any condition that would significantly affect the participant's ability to adhere to the protocol, affect interpretation of the study results, or put the participant at unacceptable risk for study-related complications as judged by the referring clinician. This may include a) patients with a specific acute contraindication to receiving ECP due to any acute condition such as new or evolving myocardial infarction or central nervous system disorder, hemodynamic instability or hypovolemia, acute bleeding, respiratory distress.
5. Patients with lupus erythematosus, porphyria cutanea tarda, erythropoietic protoporphyria, variegate porphyria, xeroderma pigmentosum, albinism, or other dermatologic or ocular condition that contraindicates the use of methoxsalen or markedly enhances photosensitivity in the investigator's judgment.
6. Aphakia or absence of ocular lenses
7. Pregnancy (positive pregnancy test - a urine or blood pregnancy test must be obtained within 2 weeks prior to enrollment in women of childbearing potential)
8. Inability to provide informed consent or to comply with study treatments or assessments (e.g. due to cognitive impairment or geographic distance)
9. Recent (i.e., within 2 weeks prior to enrollment) leukopenia (white blood cell count < 30K/cumm or 3,000/mm3/ or 3.0 109 /L)
10. Patients whose decline in lung function (FEV1) is related to either Restrictive Chronic Lung Allograft Dysfunction (CLAD) or other causes that do not represent BOS such as pneumonia, heart failure, etc.

    For patients under review for eligibility for ECP for refractory BOS:
11. Patients with a post-transplant baseline FEV1 > 3 liters and most recent FEV1 < 900 mL
12. Patients with a post-transplant FEV1< 3 liters and the most recent FEV1 < 30% of post-transplant baseline
13. Rate of FEV1 decline within the last 6 or 9 months > 300 mL/month.
14. History of receiving ECP therapy within 6 months prior to enrollment.

    For patients under review for eligibility for RCT:
15. Patients post-transplant treated with any agent that depletes T lymphocytes for In-duction, acute cellular rejection or for any other reason can only be enrolled 12 months after the last dose of these agents assuming they meet enrollment inclusion criteria. T Lymphocyte depleting therapies include (but not limited to):

    ⦁ monoclonal antibodies such as Alemtuzumab (Campath) that target CD52 T cell receptors

    ⦁ polyclonal antibodies such as anti-thymocyte globulin (ATG) via immunization of rabbits (rATG) to either human thymocytes or Jurkat cells or via immunization of horses (hATG) to human thymocytes

    ⦁ Radiation. Anti-B cell agents that do not deplete T lymphocytes such as Rituximab can be used and will not affect eligibility.
16. Any patient who at least 6 months after transplant is treated with an escalated dose of steroids (i.e., prednisone greater than 30 mg/day or that exceeds 900 mg in a 30 day period or equipotent doses of other steroids like Solumedrol ) for more than one month for an acute decline in lung function that is suspected to be secondary to acute cellular rejection.

INCLUSION CRITERIA for Refractory BOS Standard of Care Comparator using data obtained from a retrospective chart review

1. Age (18 years or older) 2. Identification of Insurance Payer (Medicare bs third party payers) 3. Lung transplant recipient (combined organ transplant recipients, e.g. heart-lung or liver- lung recipients), or lung re-transplantation are eligible) before 2022.

4. Development of BOS between 2016-2022 and was NOT treated with ECP and must be at least one year after transplant.

5. Availability of at least three spirometry values within 14 months prior to the BOS diagnosis.

EXCLUSION CRITERIA for Refractory BOS Standard of Care Comparator using data obtained from a retrospective chart review

1. Participation in a clinical treatment trial with an investigational agent used to manage BOS
2. Pregnancy
3. Patients whose decline in lung function (FEV1) is related to either Restrictive CLAD or other causes that do not represent BOS such as pneumonia, heart failure, etc.
4. History of receiving ECP Therapy for BOS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2015-01; Primary Completion 2027-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
REFRACTORY BOS: Change in the rate of FEV1 decline. | Baseline vs 12 months following the initiation of ECP.
  Comparing the average rate of FEV1 (from pulmonary function test (PFT) or spirometry) decline over the 6 months prior to ECP against the average rate of FEV1 decline over the 12 months following initiation of ECP. A clinical response will be defined as a 50% or greater reduction in the rate of decline of FEV1 before and after the ECP treatment.
NEW BOS: Cumulative All-cause mortality | 5 Years following randomization
  Survival in patients assigned to ECP treatment compared to survival in patients assigned to standard of care. A measure looking at total number of deaths from any cause.
NEW BOS: Change in the rate of FEV1 decline | Baseline vs 12 months following randomization
  A 25% or greater difference in the percentage of patients within each of the two arms (Control vs EPI) who achieve a clinical response which is defined by a 50% or greater reduction in the rate of FEV1 decline as assessed by comparing the average rate of FEV1 decline over the 6 months prior to ECP Treatment against the average rate of FEV1 decline over the 12 months following randomization.
REFRACTORY BOS: All cause and CLAD related mortality | 5 years following enrollment or the initial ECP.
  A measure looking at total number of deaths from any cause and total number of CLAD related deaths. Outcome 1 (above) and this Outcome 4 will be assessed with two comparisons as follows:(1) Comparison of the spirometric endpoint within the patients enrolled in the rBOS Arm when each patient is used as their own control. (2) The ECP Treatment Cohort (i.e., rBOS patients within the ECP Registry initially assigned to ECP treatment that have completed the six-month ECP regiment) will be compared to a propensity matched standard of care cohort based on one or more potential spirometric values (e.g. % of baseline FEV1 and possibly rate of FEV1 decline at enrollment and/or comorbidity variables at BOS diagnosis). The standard of care cohort will be captured using data obtained via a retrospective chart review at each collaborating site.

SECONDARY OUTCOMES:
All Participants: Average rate of FEV1 decline over the 9 months following initiation of ECP treatment in Refractory BOS or randomization in NEW BOS or the Randomized Control Trial. | Baseline vs 9 Months following randomization
  Look at the average rate of FEV1 decline obtained from a pulmonary function test or spirometry over the 9 months following initiation of ECP.
All Participants: All-cause and CLAD related mortality following either randomization (NEW BOS) or initiation of ECP (Refractory BOS) | Annually for five years
  A measure looking at total number of deaths from any cause and total number of CLAD related deaths.
All Participants: Proportion of patients with treatment-related serious adverse events after randomization in RCT or NEW BOS or after ECP initiation in Refractory BOS | Every 6 months for up to 5 years following enrollment.
  Review number of patients with treatment related serious adverse events in both groups.
All Participants: Change in Health-Related Quality of Life | Baseline and months 3, 6, 9, and 12, and annually up to 5 years.
  The Quality of Life Questionnaire has combined the Dyspnea 12, the Modified Medical Research Council Dyspnea Scale, The St Georges' Respiratory Questionnaire, and the EQ-5D-5L. The Dyspnea12 questionnaire assesses dyspnea severity and is comprised of 12 items and two domains (Physical: 7 questions, affective: 5 questions). Participants are instructed to indicate how much (None =0, Mild=1, Moderate=2, Severe=3) each item "troubled you". The Modified Medical Research Council Dyspnea Scale comprises 5 statements that describe the range of respiratory disability from none (Grade 0 ) to almost complete incapacity (Grade 5). The St. Georges addresses the frequency of respiratory symptoms and the patient's current state. Each question response has a unique weight. The lowest is 0 and the highest is 100. EQ-5D-5L comprises 5 dimensions: mobility, self-care, usual activities, pain and anxiety/depression. The Scores will be totaled and compared between the treatment and control group
All Participants: Effect of maintenance ECP (number of procedures and duration) on BOS progression and outcome. | At the end of 5 year follow-up
  Look at number of maintenance ECP procedures and duration of maintenance ECP treatments and its effect on BOS progression and patient's outcome.
All Participants: Diagnostic performance of our spirometric enrollment criteria | After enrollment of 80 refractory BOS patients. Will be assessed with the RCT or NEW BOS patients at the end of the study.
  Identify patients who have a response by review of rate and statistical significance of decline in FEV1. (i.e., > 50% decline in the rate of FEV1 decline).
NEW BOS: A 30% increase in residual of FEV1 values in BOS treatment Arm (EPI or Control); this would include all patients and spirometry monitoring sub-cohorts. | 6 months after randomization
  Residual FEV1 obtained at one or more post enrollment time periods is defined as any of the following values: FEV1, FEV1 as % of post-transplant baseline and FEV1 as % of enrollment FEV1.
NEW BOS: Incidence of pulmonary specific infections, CVC related infections and all infections. | 5 years
  Review of the occurrence, rate, and/or frequency of the number of pulmonary specific infections, catheter related infections and all infections in the NEW BOS group
NEW BOS: Hospitalization rates between EPI and control arms | 5 years after enrollment.
  Compare hospitalization rates between the two arms.
NEW BOS: Treatment related serious adverse events (SAEs) between EPI and control arms. | Every 6 months up to 5 years after enrollment
  Compare treatment related SAEs between early ECP treatment intervention to the control group
REFRACTORY BOS: Additional analyses will be performed to evaluate the validity of the study's FEV1-based treatment allocation method using data from enrollees in both the Observation and ECP Treatment groups | 5 years after enrollment
  How accurately did the FEV1 based treatment allocation method predict that the participant was placed in the right group i.e. ECP treatment vs observation.

CONTACTS AND LOCATIONS:
Overall Officials: George J. Despotis, M.D., Principal Investigator — Washington University St. Louis School of Medicine
Locations (22):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of California San Diego, La Jolla, California
  - University of Florida, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist, Houston, Texas
  - Inova Health System, Falls Church, Virginia

REFERENCES:
- [Background] Burton CM, Carlsen J, Mortensen J, Andersen CB, Milman N, Iversen M. Long-term survival after lung transplantation depends on development and severity of bronchiolitis obliterans syndrome. J Heart Lung Transplant. 2007 Jul;26(7):681-6. doi: 10.1016/j.healun.2007.04.004. PMID 17613397
- [Background] Hadjiliadis D, Steele MP, Govert JA, Davis RD, Palmer SM. Outcome of lung transplant patients admitted to the medical ICU. Chest. 2004 Mar;125(3):1040-5. doi: 10.1378/chest.125.3.1040. PMID 15006966
- [Background] Morrell MR, Despotis GJ, Lublin DM, Patterson GA, Trulock EP, Hachem RR. The efficacy of photopheresis for bronchiolitis obliterans syndrome after lung transplantation. J Heart Lung Transplant. 2010 Apr;29(4):424-31. doi: 10.1016/j.healun.2009.08.029. Epub 2009 Oct 22. PMID 19853479
- [Result] Reviewed in: Centers for Medicare and Medicaid Services. Final Decision Memorandum for Extracorporeal Photophresis (CAG-00324R), April 2012
- [Derived] Chionis L, Grossman BJ, Hachem R, Commean P, Derfler MC, Vedantham S, Dodds K, Spitznagel E, Atkinson J, Despotis G. The efficacy of extracorporeal photopheresis to arrest bronchiolitis obliterans in lung allograft recipients was compared between two automated photopheresis instruments. Transfusion. 2018 Dec;58(12):2933-2941. doi: 10.1111/trf.14913. Epub 2018 Oct 12. PMID 30312482